CLINICAL TRIAL: NCT00457743
Title: A Phase I/II Study of Sunitinib Malate (SU011248) In The Treatment of Patients With Malignant Gastrointestinal Stromal Tumor (GIST) Previously Treated by Imatinib Mesylate.
Brief Title: A Phase I/II Study of Sunitinib Malate (SU011248) In Patients With Gastrointestinal Stromal Tumor (GIST)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181045; JapicCTI-070386
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-10

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Evaluate of RTD for Japanese GIST patients
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SU011248 (Experimental): 25 , 50 or 75 mg/day of SU011248
  Interventions: Drug: Sunitinib malate (SU011248)

INTERVENTIONS:
Drug: Sunitinib malate (SU011248) — SU011248

SUMMARY:
Phase I;To investigate the clinically recommended dose of Sunitinib malate (SU011248) following multiple oral dosing in the first cycle (4 consecutive weeks and 2 weeks rest) by reviewing the safety and tolerability.

Phase II;To determine the objective tumor response and the safety of Sunitinib malate (SU011248) at the clinically recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed metastatic or unresectable gastrointestinal stromal tumor (GIST).
* Patients previously treated with imatinib mesylate.

Exclusion Criteria:

* Patients who have not recovered from the acute toxic effects of previous antineoplastic therapy or treatment with imatinib mesylate.
* Any tumor therapy for gastrointestinal stromal tumor (GIST) discontinued less than 4 weeks prior to starting study treatment. Imatinib mesylate discontinued less than 2 weeks prior to starting therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Pfizer Investigational Site, Kashiwa, Chiba
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Suita, Osaka
  - Pfizer Investigational Site, Chuo-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181045&StudyName=A%20Phase%20I/II%20Study%20of%20%20Sunitinib%20malate%20%28SU011248%29%20In%20Patients%20with%20Gastrointestinal%20Stromal%20Tumor%20%28GIST%29%20%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1 only included Cycle 1 for subjects enrolled in Phase 1. Phase 2 was comprised of either Cycle 2 and beyond for subjects who were enrolled in Phase 1, or all cycles for newly enrolled subjects. Additional subjects were enrolled to make a total of 30 in the recommended dose level (50-mg).
Groups:
- SU-011248 25-mg: Subjects received sunitinib malate (SU-011248) at starting dose of 25-mg once daily. Treatment cycles were 6 weeks in duration, consisting of 4 weeks daily SU-011248 administration followed by 2 weeks off treatment.
  Phase 1: If Dose Limiting Toxicity (DLT) was observed, the patients were withdrawn from the study treatment. Neither temporary discontinuation nor reduction was permitted.
  Phase 2: The initial dose could be increased to the recommended dose. Treatment cycles were repeated until a study treatment withdrawal criterion was met. If drug-related adverse event (grade>=3) was observed, temporary discontinuation or dose reduction were taken according to the criteria.
- SU-011248 50-mg: Subjects received sunitinib malate (SU-011248) at starting dose of 50-mg once daily. Treatment cycles were 6 weeks in duration, consisting of 4 weeks daily SU-011248 administration followed by 2 weeks off treatment.
  Phase 1: If Dose Limiting Toxicity (DLT) was observed, the patients were withdrawn from the study treatment. Neither temporary discontinuation nor reduction was permitted.
  Phase 2: Treatment cycles were repeated until a study treatment withdrawal criterion was met. If drug-related adverse event (grade>=3) was observed, temporary discontinuation or dose reduction were taken according to the criteria.
  From Phase 1 part of this study, 50-mg was determined as the maximum tolerated dose and the recommended dose.
- SU-011248 75-mg: Subjects received sunitinib malate (SU-011248) at starting dose of 75-mg once daily. Treatment cycles were 6 weeks in duration, consisting of 4 weeks daily SU-011248 administration followed by 2 weeks off treatment.
  Phase 1: If Dose Limiting Toxicity (DLT) was observed, the patients were withdrawn from the study treatment. Neither temporary discontinuation nor reduction was permitted.
  Phase 2: The initial dose could be reduced to the recommended dose. Treatment cycles were repeated until a study treatment withdrawal criterion was met. If drug-related adverse event (grade>=3) was observed, temporary discontinuation or dose reduction were taken according to the criteria.
Period: Overall Study
Arm/Group | SU-011248 25-mg | SU-011248 50-mg | SU-011248 75-mg
Started | 3 (Overall study) | 30 (Overall study) | 3 (Overall study)
Enrolled in Phase 1 | 3 | 6 | 3
Completed Phase 1 | 3 | 6 | 3
Enrolled in Phase 2 | 3 (Three subjects who completed Phase 1 entered Phase 2.) | 30 (Six subjects who completed Phase 1 entered Phase 2, and 24 subjects were newly enrolled.) | 3 (Three subjects who completed Phase 1 entered Phase 2.)
Completed | 0 (However, all 3 subjects enrolled were included in analysis (Intent-to treat population).) | 3 (However, all 30 subjects enrolled were included in analysis(Intent-to treat population).) | 0 (However, all 3 subjects enrolled were included in analysis(Intent-to treat population).)
Not Completed | 3 | 27 | 3
Not completed — Adverse Event | 0 | 4 | 0
Not completed — Lack of Efficacy | 3 | 23 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SU-011248 25-mg | SU-011248 50-mg | SU-011248 75-mg | Total
Number analyzed (Participants) | 3 | 30 | 3 | 36
Age, Customized [Number; unit: participants]
  18-44 years | 2 | 2 | 0 | 4
  45-64 years | 1 | 24 | 1 | 26
  >=65 years | 0 | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 0 | 12
  Male | 2 | 19 | 3 | 24
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 30 | 3 | 36
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  participants
    0 | 3 | 18 | 2 | 23
    1 | 0 | 12 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLT)
Description: Dose Limiting Toxicities(DLT) in the subjects enrolled in Phase 1.
Time Frame: Cycle 1 (Baseline to Week 6)
Population: DLT analysis population consists of subjects who developed DLT or received 85% of the planned dose. One subject in 75-mg dose group was excluded from DLT analysis population because the subject received less than 85% of the planned dose.
Measure: Number; unit: participants
Arm/Group | SU-011248 25-mg | SU-011248 50-mg | SU-011248 75-mg
Number analyzed (Participants) | 3 | 6 | 2
participants | 0 | 0 | 2

2. Primary Outcome: Maximum Plasma Concentration (Cmax) on Cycle 1 Day 1
Description: Maximum Plasma Concentration (Cmax) of SU-011248, its active metabolite SU-012662 and Total drug (SU-011248+SU-012662) in the subjects enrolled in Phase 1.
  The Cmax for total drug (SU-011248+SU-012662) was calculated as the mean of the Cmax of total drug from each individual subject (it is not the simple sum of means of Cmax of SU-011248 and SU-012662).
Time Frame: Day 1 of Cycle 1
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 blood concentration data for Pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU-011248 25-mg | SU-011248 50-mg | SU-011248 75-mg
Number analyzed (Participants) | 3 | 6 | 3
ng/mL
  SU-011248 | 12.1 (4.9) | 22.8 (6.4) | 32.3 (20.8)
  SU-012662 | 1.96 (1.27) | 4.13 (0.93) | 4.81 (2.54)
  SU-011248+SU-012662 | 14.1 (6.1) | 26.7 (7.4) | 37.0 (22.1)

3. Secondary Outcome: Plasma Concentrations of Vascular Endothelial Growth Factor (VEGF)
Description: Plasma concentrations of potential pharmacodynamic markers; Vascular Endothelial Growth Factor (VEGF)
Time Frame: Day 1, 14, 28 of Cycles 1-4
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 blood concentration data for Pharmacodynamics analysis.
  n= Number of subjects with analyzable data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
pg/mL
  Cycle 1 Day 1 (n=30) | 55.30 (32.43)
  Cycle 1 Day 14 (n=30) | 179.94 (116.00)
  Cycle 1 Day 28 (n=19) | 192.42 (210.58)
  Cycle 2 Day 1 (n=26) | 62.05 (38.20)
  Cycle 2 Day 14 (n=24) | 173.12 (96.30)
  Cycle 2 Day 28 (n=20) | 207.79 (158.05)
  Cycle 3 Day 1 (n=18) | 58.80 (26.13)
  Cycle 3 Day 14 (n=19) | 208.93 (159.41)
  Cycle 3 Day 28 (n=13) | 238.74 (227.63)
  Cycle 4 Day 1 (n=11) | 54.83 (14.86)
  Cycle 4 Day 14 (n=12) | 227.28 (163.52)
  Cycle 4 Day 28 (n=9) | 343.21 (210.28)

4. Secondary Outcome: Plasma Concentrations of Soluble Vascular Endothelial Growth Factor Type 2 Receptors (sVEGFR2)
Description: Plasma concentrations of potential pharmacodynamic markers; Soluble Vascular Endothelial Growth Factor Type 2 Receptors (sVEGFR2)
Time Frame: Day 1, 14, 28 of Cycles 1-4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
pg/mL
  Cycle 1 Day 1 (n=30) | 8740.20 (1702.84)
  Cycle 1 Day 14 (n=30) | 5721.98 (1136.89)
  Cycle 1 Day 28 (n=19) | 5082.92 (1449.26)
  Cycle 2 Day 1 (n=26) | 7579.98 (1844.58)
  Cycle 2 Day 14 (n=24) | 5808.08 (1484.30)
  Cycle 2 Day 28 (n=20) | 4770.15 (1311.88)
  Cycle 3 Day 1 (n=18) | 6802.86 (1641.46)
  Cycle 3 Day 14 (n=19) | 5022.84 (1192.52)
  Cycle 3 Day 28 (n=13) | 4297.91 (1157.62)
  Cycle 4 Day 1 (n=11) | 6559.50 (1152.24)
  Cycle 4 Day 14 (n=12) | 5038.50 (1078.45)
  Cycle 4 Day 28 (n=9) | 4142.72 (1103.29)

5. Secondary Outcome: Plasma Concentrations of Soluble Stem Cell Factor Receptor (sKIT)
Description: Plasma concentrations of potential pharmacodynamic markers; Soluble Stem Cell Factor Receptor (sKIT)
Time Frame: Day 1, 14, 28 of Cycles 1-4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
pg/mL
  Cycle 1 Day 1 (n=30) | 48237.33 (56643.93)
  Cycle 1 Day 14 (n=30) | 53087.75 (71243.85)
  Cycle 1 Day 28 (n=19) | 35538.95 (16082.33)
  Cycle 2 Day 1 (n=26) | 39011.35 (38304.60)
  Cycle 2 Day 14 (n=24) | 40432.29 (45085.57)
  Cycle 2 Day 28 (n=20) | 30715.75 (16212.04)
  Cycle 3 Day 1 (n=18) | 27814.17 (10362.85)
  Cycle 3 Day 14 (n=19) | 32973.68 (14483.42)
  Cycle 3 Day 28 (n=13) | 32760.77 (16888.75)
  Cycle 4 Day 1 (n=11) | 28961.82 (14899.42)
  Cycle 4 Day 14 (n=12) | 32265.83 (16143.54)
  Cycle 4 Day 28 (n=9) | 32571.11 (20949.63)

6. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-011248
Description: Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration
Time Frame: Day 14, 28 of Cycle 1; Day 1, 14, 28 of Cycles 2-4
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 blood concentration data for Pharmacokinetic analysis.
  n= Number of subjects with analyzable data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
ng/mL
  Cycle 1 Day 14 (n=28) | 58.93 (23.87)
  Cycle 1 Day 28 (n=18) | 44.52 (15.45)
  Cycle 2 Day 1 (n=15) | 1.17 (0.60)
  Cycle 2 Day 14 (n=23) | 51.23 (16.98)
  Cycle 2 Day 28 (n=20) | 48.09 (22.41)
  Cycle 3 Day 1 (n=11) | 1.62 (0.88)
  Cycle 3 Day 14 (n=14) | 58.72 (27.09)
  Cycle 3 Day 28 (n=10) | 47.13 (21.73)
  Cycle 4 Day 1 (n=5) | 1.52 (0.81)
  Cycle 4 Day 14 (n=7) | 46.13 (22.28)
  Cycle 4 Day 28 (n=8) | 47.33 (12.95)

7. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-012262
Description: Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration
Time Frame: Day 14, 28 of Cycle 1; Day 1, 14, 28 of Cycles 2-4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
ng/mL
  Cycle 1 Day 14 (n=28) | 26.41 (15.86)
  Cycle 1 Day 28 (n=18) | 24.52 (13.28)
  Cycle 2 Day 1 (n=15) | 2.01 (0.90)
  Cycle 2 Day 14 (n=23) | 24.06 (11.54)
  Cycle 2 Day 28 (n=20) | 24.47 (14.92)
  Cycle 3 Day 1 (n=11) | 2.26 (1.20)
  Cycle 3 Day 14 (n=14) | 27.69 (16.34)
  Cycle 3 Day 28 (n=10) | 23.83 (12.59)
  Cycle 4 Day 1 (n=5) | 2.02 (0.90)
  Cycle 4 Day 14 (n=7) | 19.86 (11.38)
  Cycle 4 Day 28 (n=8) | 25.94 (12.28)

8. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-011248+SU-012662
Description: Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration
Time Frame: Day 14, 28 of Cycle 1; Day 1, 14, 28 of Cycles 2-4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
ng/mL
  Cycle 1 Day 14 (n=28) | 85.33 (36.59)
  Cycle 1 Day 28 (n=18) | 69.05 (27.52)
  Cycle 2 Day 1 (n=15) | 3.18 (1.45)
  Cycle 2 Day 14 (n=23) | 75.29 (27.35)
  Cycle 2 Day 28 (n=20) | 72.56 (36.14)
  Cycle 3 Day 1 (n=11) | 3.88 (1.88)
  Cycle 3 Day 14 (n=14) | 86.41 (42.83)
  Cycle 3 Day 28 (n=10) | 70.96 (32.81)
  Cycle 4 Day 1 (n=5) | 3.54 (1.46)
  Cycle 4 Day 14 (n=7) | 65.99 (33.42)
  Cycle 4 Day 28 (n=8) | 73.26 (24.82)

9. Secondary Outcome: Changes From Baseline of Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Questionnaires
Description: Patient-reported outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) questionnaires (version 4A).
  The questionnaire consists of a 13-item subscale which covers specific fatigue questions. The subject rates the intensity of fatigue and its related symptoms on a five-point scale(0 to 4). High score is indicating low fatigue. The total score of the 13 items was evaluated.
  Change from Baseline: Score at each observation minus score at baseline
Time Frame: Day 7, 14, 28, 35 of Cycle 1; Day 1, 7, 14, 28, 35 of Cycles 2-4
Population: Intent-to-Treat (ITT) population defined as all subjects enrolled in study that receive at least 1 dose of study medication.
  n= Number of subjects with analyzable data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
scores on a scale
  Cycle 1 Day 7 (n=30) | 1.0 (5.6)
  Cycle 1 Day 14 (n=30) | -2.3 (7.8)
  Cycle 1 Day 21 (n=30) | -6.3 (13.8)
  Cycle 1 Day 28 (n=30) | -4.6 (10.2)
  Cycle 1 Day 35 (n=30) | -0.4 (6.6)
  Cycle 2 Day 1 (n=30) | 1.5 (5.8)
  Cycle 2 Day 7 (n=30) | -0.2 (8.0)
  Cycle 2 Day 14 (n=30) | -1.3 (8.7)
  Cycle 2 Day 21 (n=30) | -3.6 (10.5)
  Cycle 2 Day 28 (n=29) | -5.1 (10.6)
  Cycle 2 Day 35 (n=29) | -2.5 (8.7)
  Cycle 3 Day 1 (n=25) | -1.3 (8.6)
  Cycle 3 Day 7 (n=24) | -1.2 (6.6)
  Cycle 3 Day 14 (n=25) | -1.8 (9.3)
  Cycle 3 Day 21 (n=24) | -4.8 (9.8)
  Cycle 3 Day 28 (n=25) | -3.8 (10.0)
  Cycle 3 Day 35 (n=25) | -3.4 (10.4)
  Cycle 4 Day 1 (n=21) | -2.7 (9.5)
  Cycle 4 Day 7 (n=20) | -4.4 (11.4)
  Cycle 4 Day 14 (n=21) | -6.2 (11.5)
  Cycle 4 Day 21 (n=20) | -8.8 (12.5)
  Cycle 4 Day 28 (n=19) | -9.7 (11.5)
  Cycle 4 Day 35 (n=20) | -8.6 (11.2)

10. Secondary Outcome: Change From Baseline of European Quality of Life Questionnaire- 5 Dimensions(EQ-5D) Questionnaires
Description: The EQ-5D questionnaires evaluates 5 dimensions of health. The subjects rates the severity of impairment for each dimensions on a 3-point scale(1 to 3). The digits for five dimensions were combined in a five-digit number describing the respondent's health state. Health states were converted into a weighted health state index. High score is indicating high health.
  Change from Baseline: weighted health state index at each observation minus weighted health state index at baseline
Time Frame: Day 28 of Cycle 1; Day 1, 28 of Cycles 2-4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: index scores on a scale
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
index scores on a scale
  Cycle 1 Day 28 (n=30) | -0.148 (0.213)
  Cycle 2 Day 1 (n=30) | -0.038 (0.171)
  Cycle 2 Day 28 (n=30) | -0.121 (0.215)
  Cycle 3 Day 1 (n=25) | -0.010 (0.125)
  Cycle 3 Day 28 (n=25) | -0.091 (0.210)
  Cycle 4 Day 1 (n=21) | -0.006 (0.137)
  Cycle 4 Day 28 (n=18) | -0.142 (0.198)

11. Secondary Outcome: Number of Subjects With Disease Controlled Based on the Extramural Review Committee Assessment in Recommended Dose Group
Description: Number of subjects with Disease Controlled is defined as sum of the subjects confirmed with complete response (CR), partial response (PR), or stable disease (SD)>= 10 weeks on study according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Day 28 of Cycles 1-4
Population: Intent-to-Treat (ITT) population defined as all subjects enrolled in study that receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
participants
  Total number of Subjects with CR+PR+SD>=10weeks | 17
  Complete Response (CR) | 0
  Partial Response (PR) | 4
  Stable Disease (SD) >= 10 weeks | 13
Statistical Analysis 1: Comparison: SU-011248 50-mg; Test type: Superiority or Other; Disease control Rate (percentage) = 56.7, 95% CI [37.4 to 74.5] — The disease control rate, defined as the percentage of subjects confirmed with CR, PR, and SD >=10 weeks on study according to RECIST

12. Primary Outcome: Maximum Plasma Concentration (Cmax) on Cycle 1 Day 28
Description: as for outcome 2
Time Frame: Day 28 of Cycle 1
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 blood concentration data for Pharmacokinetic analysis.
  3 subjects in 75mg dose group discontinued before Cycle 1 Day 28, therefore no data presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU-011248 25-mg | SU-011248 50-mg
Number analyzed (Participants) | 3 | 6
ng/mL
  SU-011248 | 39.5 (25.0) | 69.3 (18.9)
  SU-012662 | 15.2 (10.2) | 38.8 (16.0)
  SU-011248+SU-012662 | 54.0 (32.2) | 105 (35)

13. Secondary Outcome: Number of Subjects With Objective Response Based on the Extramural Review Committee Assessment in Recommended Dose Group
Description: Number of subjects with Objective Response is defined as sum of the subjects confirmed with complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Day 28 of Cycles 1-4
Population: ITT population defined as all subjects enrolled in study that receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
participants
  Total Number of Subjects with CR+PR | 4
  Complete Response (CR) | 0
  Partial Response (PR) | 4
Statistical Analysis 1: Comparison: SU-011248 50-mg; Test type: Superiority or Other; Objective Response Rate(percentage) = 13.3, 95% CI [3.8 to 30.7] — The subjects confirmed with complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST)

14. Secondary Outcome: Time To Tumor Progression (TTP)
Description: Time To tumor Progression (TTP) is defined as the time from the date of first dose of study treatment to the date of the first documentation of Progressive Disease (PD).
Time Frame: From the first dose to Progressive Disease
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
Weeks | 30.3 [22.0 to 46.1]

15. Primary Outcome: Area Under the Plasma Concentration Curve (AUC0-24) on Cycle 1 Day 1
Description: Area Under the Plasma Concentration Curve (AUC0-24) of SU-011248, its active metabolite SU-012662 and Total drug (SU-011248+SU-012662) in the subjects enrolled in Phase 1.
  The AUC0-24 for total drug (SU-011248+SU-012662) was calculated as the mean of the AUC0-24 of total drug from each individual subject (it is not the simple sum of means of AUC0-24 of SU-011248 and SU-012662).
Time Frame: Day 1 of Cycle 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | SU-011248 25-mg | SU-011248 50-mg | SU-011248 75-mg
Number analyzed (Participants) | 3 | 6 | 3
ng•h/mL
  SU-011248 | 199 (89) | 374 (69) | 508 (259)
  SU-012662 | 30.9 (20.6) | 70.0 (14.4) | 91.1 (45.3)
  SU-011248+SU-012662 | 230 (108) | 444 (82) | 599 (287)

16. Primary Outcome: Area Under the Plasma Concentration Curve (AUC0-24) on Cycle 1 Day 28
Description: as for outcome 15
Time Frame: Day 28 of Cycle 1
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 blood concentration data for Pharmacokinetic analysis.
  3 subjects in 75-mg dose group discontinued the dose on Cycle1, therefore no data showed.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | SU-011248 25-mg | SU-011248 50-mg
Number analyzed (Participants) | 3 | 6
ng•h/mL
  SU-011248 | 858 (600) | 1406 (364)
  SU-012662 | 324 (223) | 772 (358)
  SU-011248+SU-012662 | 1182 (734) | 2178 (702)

17. Primary Outcome: Time to First Occurrence of Cmax (Tmax) on Cycle 1 Day 1
Description: Time to First Occurrence of Cmax (Tmax) of SU-011248, its active metabolite SU-012662 and Total drug (SU-011248+SU-012662) in the subjects enrolled in Phase 1.
  The Tmax for total drug (SU-011248+SU-012662) was calculated as the median of the Tmax of total drug from each individual subject (it is not the simple sum of median of Tmax of SU-011248 and SU-012662).
Time Frame: Day 1 of Cycle 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | SU-011248 25-mg | SU-011248 50-mg | SU-011248 75-mg
Number analyzed (Participants) | 3 | 6 | 3
hours
  SU-011248 | 6 [4 to 8] | 7 [6 to 24] | 8 [4 to 10]
  SU-012662 | 6 [4 to 8] | 9 [6 to 24] | 10 [4 to 10]
  SU-011248+SU-012662 | 6 [4 to 8] | 7 [6 to 24] | 8 [4 to 10]

18. Primary Outcome: Time to First Occurrence of Cmax (Tmax) on Cycle 1 Day 28
Description: Time to First Occurrence of Cmax (Tmax) of SU-011248, its active metabolite SU-012662 and Total drug (SU-011248+SU-012662) in the subjects enrolled in Phase 1.
  The Tmax for total drug (SU-011248+SU-012662) was calculated as the median of the Tmax of total drug from each individual subject (it is not the simple sum of medians of Tmax of SU-011248 and SU-012662).
Time Frame: Day 28 of Cycle 1
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 blood concentration data for Pharmacokinetic analysis.
  3 subjects in 75-mg dose group discontinued before Cycle 1 Day 28, therefore no data presented.
Measure: Median (Full Range); unit: hours
Arm/Group | SU-011248 25-mg | SU-011248 50-mg
Number analyzed (Participants) | 3 | 6
hours
  SU-011248 | 10 [6 to 10] | 6 [1 to 24]
  SU-012662 | 4 [2 to 8] | 2.5 [0 to 48]
  SU-011248+SU-012662 | 6 [4 to 8] | 6 [0 to 24]

19. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from the date of first dose of study treatment to the date of the first documentation of Progressive Disease (PD) or death.
Time Frame: From the first dose to Progressive Disease or Death
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
Weeks | 30.3 [22.0 to 46.1]

20. Primary Outcome: SU-011248 Clearance on Cycle 1 Day 28
Description: SU-011248 Clearance in the subjects enrolled in Phase 1.
  Clearance was calculated by dividing a SU-011248 dose(mg) by AUC0-24(ng•h/mL).
Time Frame: Day 28 of Cycle 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | SU-011248 25-mg | SU-011248 50-mg
Number analyzed (Participants) | 3 | 6
L/h | 43.1 (32.8) | 38.1 (11.6)

21. Primary Outcome: Accumulation Ratio (Rac) on Cycle 1 Day 28
Description: Accumulation Ratio (Rac) of SU-011248, its active metabolite SU-012662 and Total drug (SU-011248+SU-012662) on Cycle 1 Day 28 in the subjects enrolled in Phase 1.
  Rac was the ratio of Day 28 to Day 1.
Time Frame: Day 28 of Cycle 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | SU-011248 25-mg | SU-011248 50-mg
Number analyzed (Participants) | 3 | 6
ratio
  SU-011248: Rac Cmax | 3.32 (2.17) | 3.10 (0.77)
  SU-011248: Rac AUC0-24 | 4.31 (2.65) | 3.76 (0.82)
  SU-012662: Rac Cmax | 7.98 (4.91) | 9.00 (2.20)
  SU-012662: Rac AUC0-24 | 10.4 (5.5) | 10.6 (3.5)
  SU-011248+SU-012662: Rac Cmax | 3.87 (2.36) | 3.93 (0.98)
  SU-011248+SU-012662: Rac AUC0-24 | 5.08 (2.74) | 4.85 (1.20)

22. Primary Outcome: Number of Subjects With Clinical Benefit Response (CBR) Based on the Extramural Review Committee Assessment in Recommended Dose Group
Description: Clinical Benefit Response is defined as sum of subjects confirmed with complete response (CR), partial response (PR), or stable disease (SD)>= 22 weeks on study according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Day 28 of Cycles 1-4
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
participants
  Total Number of Subjects with CR+PR+SD>=22weeks | 12
  Complete Response (CR) | 0
  Partial Response (PR) | 4
  Stable Disease (SD) >= 22 weeks | 8
Statistical Analysis 1: Comparison: SU-011248 50-mg; Test type: Superiority or Other; CBR rate (percentage) = 40.0, 95% CI [22.7 to 59.4] — The clinical benefit response (CBR) rate, defined as the percentage of the subjects confirmed with CR, PR, or SD>=22 weeks on study according to Response Evaluation Criteria in Solid Tumors (RECIST)

23. Secondary Outcome: Time To Failure (TTF)
Description: Time To Failure (TTF) is defined as the time from the date of first dose of study treatment to the date of the first documentation of Progressive Disease (PD), the date of treatment discontinuation except completion of treatment, or date of death due to cancer.
Time Frame: From the first dose to Progressive Disease, Treatment discontinuation except completion of treatment, or Death due to cancer.
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
Weeks | 28.4 [21.9 to 46.1]

24. Secondary Outcome: Overall Survival Time
Description: Overall Survival Time is defined as the time from the date of first dose of study treatment to the date of the death due to any cause. For subjects whose death had not been confirmed, Overall Survival Time was censored on the last date when the patient was known to be alive.
  Survival was surveyed once a year from the registration day of the first subject, for all the subjects who received the study drug at least once.
Time Frame: From the first dose to death
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | SU-011248 50-mg
Number analyzed (Participants) | 30
Weeks | 62.0 [47.9 to 99.9]

ADVERSE EVENTS:
Arm/Group | SU-011248 25-mg | SU-011248 50-mg | SU-011248 75-mg
Serious Adverse Events (participants affected / at risk) | 1/3 | 12/30 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 30/30 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SU-011248 25-mg (N=3) | SU-011248 50-mg (N=30) | SU-011248 75-mg (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SU-011248 25-mg (N=3) | SU-011248 50-mg (N=30) | SU-011248 75-mg (N=3)
Abdominal distension (Gastrointestinal disorders) | 1 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 17 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 14 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 22 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 18 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1
Blood albumin decreased (Investigations) | 0 | 17 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 11 | 3
Blood amylase increased (Investigations) | 0 | 8 | 3
Blood bilirubin increased (Investigations) | 1 | 9 | 2
Blood calcium decreased (Investigations) | 0 | 4 | 1
Blood creatinine increased (Investigations) | 1 | 10 | 1
Blood glucose increased (Investigations) | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 12 | 2
Blood phosphorus decreased (Investigations) | 0 | 3 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 1 | 2
Blood urea increased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 3 | 0
C-reactive protein increased (Investigations) | 0 | 4 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 9 | 1
Chest pain (General disorders) | 1 | 2 | 0
Chills (General disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 23 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 13 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 6 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Eyelid oedema (Eye disorders) | 1 | 1 | 0
Face oedema (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 2 | 23 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 13 | 0
Glossitis (Gastrointestinal disorders) | 0 | 2 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 22 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 3
Headache (Nervous system disorders) | 1 | 8 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 15 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 5 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 2 | 0
Leucine aminopeptidase increased (Investigations) | 0 | 2 | 0
Lipase increased (Investigations) | 0 | 11 | 2
Lymphocyte count decreased (Investigations) | 2 | 17 | 2
Malaise (General disorders) | 1 | 1 | 0
Monocyte count decreased (Investigations) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 10 | 1
Nausea (Gastrointestinal disorders) | 2 | 15 | 3
Nephrotic syndrome (Renal and urinary disorders) | 0 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 28 | 3
Oedema (General disorders) | 0 | 9 | 1
Oedema peripheral (General disorders) | 0 | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 26 | 3
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 3 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 9 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 7 | 2
Platelet count decreased (Investigations) | 2 | 26 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Protein total decreased (Investigations) | 0 | 8 | 2
Protein urine (Investigations) | 0 | 4 | 0
Protein urine present (Investigations) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 10 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 14 | 2
Red blood cell count decreased (Investigations) | 0 | 4 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 21 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 19 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 10 | 1
Weight decreased (Investigations) | 0 | 2 | 0
Weight increased (Investigations) | 0 | 4 | 0
White blood cell count decreased (Investigations) | 3 | 27 | 3
White blood cell count increased (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.